CLINICAL TRIAL: NCT00271258
Title: STUDY OF THE TOLERANCE OF SODIUM DIVALPROATE (DEPAKOTE) IN ADOLESCENTS IN MANIC, MIXED OR HYPOMANIC EPISODES OF BIPOLAR DISORDER
Brief Title: Safety Study of Sodium Divalproate in Bipolar Disorder in Adolescents
Acronym: ADOKOT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: L_9524; EudraCT #: 2004-004687-76
Record Dates: First submitted 2005-12-29; First posted 2005-12-30 (Estimated); Last update posted 2011-01-11 (Estimated); Status verified 2011-01

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: SODIUM DIVALPROATE

SUMMARY:
- Main objective: To evaluate the clinical and physiological tolerance of sodium divalproate in manic, mixed or hypomanic episodes of bipolar disorder in adolescents treated for 6 months.

- Secondary objective: To evaluate the efficacy of sodium divalproate in improving manic, mixed or hypomanic symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent boys or girls aged 13 to 18 inclusive
* Weighing more than 40 kg
* Capable of understanding the protocol
* Who have given their written consent, as have their parents or legal guardian unless the adolescent has passed his/her 18th birthday
* Presenting the diagnostic characteristics of manic, mixed or hypomanic episodes of bipolar disorder established in accordance with the DSM IV, gathered in a semi-structured interview (Mini International Neuropsychiatric Interview - M.I.N.I.)
* With a score on the YMRS scale (Young Mania Rating Scale) >= 14 for the manic or mixed episode or >= 10 for the hypomanic episode
* Absence in blood of valproic acid at the inclusion visit
* Willing to use effective contraception in the case of girls of child-bearing potential. In this case the investigator should satisfy him/herself as to the psychological capacity of the patient to understand and undertake use of this contraception.
* Whose physiological test results are normal: hepatic function, blood count, lipid levels, fasting blood glucose level, blood urea, blood ammonia, blood protein, serum creatinine levels and plasma ions

Exclusion Criteria:

* General criteria:

  * Pregnant girls, or those breast-feeding or those for whom a pregnancy test is positive (blood beta HCG test)
  * Simultaneous participation in another study or in the 2 months preceding selection of the patient
* Psychiatric criteria:

  * Established or known mental retardation
  * Autistic disorders
  * Established schizophrenia
  * Schizoaffective disorders
* Somatic criteria:

  * Medical or organic disease of the CNS (epilepsy, tumour etc.)
  * Any known renal, cardiac or haematological disease, or disease of the immune system
  * Endocrine disorders and/or any biochemical abnormality known or existing at the moment of inclusion
* Exclusion criteria linked to the treatment

  * Known hypersensitivity to valproate or to sodium divalproate or to one of the constituents of the drug
  * Hepatic disease: acute hepatitis, chronic hepatitis, past personal or family history of severe hepatitis particularly caused by medicinal products, hepatic porphyria
  * Treatment with lamotrigine, (Lamictal)
  * Treatment with mefloquine, (Lariam)
  * Any treatment based on valproate
  * Treatment with methylphenidate (Ritalin)

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200
Dates: Start 2005-01; Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
clinical examination

CONTACTS AND LOCATIONS:
Overall Officials: Marie SEBILLE, Dr, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Paris, France